CLINICAL TRIAL: NCT04473976
Title: Plasma Levels of CGRP and Expression of Specific microRNAs in Blood Cells of Episodic and Chronic Migraine Subjects: Toward the Identification of a Panel of Peripheral Biomarkers of Migraine?
Brief Title: Plasma Levels of CGRP and Expression of Specific microRNAs in Blood Cells of Episodic and Chronic Migraine Subjects
Acronym: CGRP-RNA
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: University of Pavia (Other)
Responsible Party: Sponsor
Other Study IDs: CGRP-microRNA2020
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Migraine
Keywords: Migraine; CGRP; MicroRNA; Overuse of medications
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples from the cubital vein of each patient was put into a 5 ml lavender tube. Plasma samples were prepared by centrifugation and then stored at -80°C. Plasma CGRP levels were measured using a commercial enzyme-linked immuno-sorbent assay kit.
  The miRNAs expression was evaluated by real-time reverse transcription (RT) Polymerase Chain Reaction (PCR) in peripheral blood mononuclear cell (PBMCs). PBMCs were isolated immediately after blood collection. Blood samples were collected within ethylenediamine tetra-acetic acid (EDTA) containing tube and diluted in 1:1 ratio with Phosphate Buffer Saline (PBS). Then, diluted blood samples were slowly loaded into Ficoll separating solution (15 ml) (Sigma) and centrifuged at 800 g for 30 min at room temperature. PBMCs accumulated as the middle white monolayer, were washed twice in sterile PBS at 300 g for 15 min. After washing, PBMCs pellet was resuspended in trizol and stored at -80 °C until use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Migraine can manifest with an episodic or chronic pattern in a continuum of disease severity. Multiple factors are associated to the transformation of the pattern form episodic to chronic. Of these, the most consistently reported is the overuse of medications (MO) for the acute treatment of attacks. Knowledge of the mechanisms through which MO facilitates the transformation of episodic migraine (EM) into chronic migraine (CM) is very limited. In order insights into these mechanisms, the present study was aimed at identifying possible peripheral biomarkers associated to the 2 forms of migraine and to the presence of MO.

The investigators evaluated CGRP plasma levels and the expression of miR-34a-5p and miR-382-5p in peripheral blood mononuclear cells of subjects with episodic migraine (EM, n=27) and CM-MO (n=28). CM-MO group was also tested 2 months after an in-hospital detoxification protocol.

DETAILED DESCRIPTION:
Chronic migraine (CM) is a highly disabling condition that frequently manifests as a negative evolution of episodic migraine (EM) taking place over years. In a recent meta-analysis on the predictors of migraine chronification, a number of monthly headache days >10 showed the strongest level of evidence, with depression and low household income being supported by moderate evidence. In the same meta-analysis, medication overuse (MO) was associated to the highest risk ratio in a random-effects model (RR 8.82; 95% Confidence Interval (CI), 2.88-27) but the strength of evidence was rated 'very low'due to substantial heterogeneity among studies.

It is likely that CM is the result of the dynamic interaction of multiple co-factors acting on a substrate represented by a more aggressive type of migraine. This hypothesis would explain why as many as 75% of CM subjects can spontaneously fluctuate around chronicity and episodicity. On the other hand, multiple pieces of evidence show that withdrawal from overuse medications induces a clinically meaningful improvement in a large percentage of subjects, with rates of benefit that are too high to be ascribed to a simple placebo effect.

The mechanisms underlying the negative effect of MO in migraine outcome are largely unknown. Neural mechanisms including a combination of nociceptive facilitation with weakened descending pain inhibition, associated with trigeminal hyperexcitability, may be involved. The loss of diffuse descending inhibition has been demonstrated in a preclinical model of CM with MO. In this frame, it is worth noting that the investigators have recently reported a marked derangement of the endocannabinoid system in subjects with CM and MO (CM-MO), which was more marked when compared with subjects suffering from episodic migraine (EM). Interestingly, detoxification induced in CM-MO subjects the normalization of pain thresholds paralleled by the reduction in headache frequency. Pre-clinical studies show that triptans, the specific symptomatic migraine drugs, induce a condition of hyperalgesia when administered chronically. Thus, it is possible that acute migraine medications taken in repeated episodes of pain may amplify the consequences of nociceptor activation and increase the probability of subsequent migraine attacks, together with the risk of medication overuse.

In this context of multiple concurrent causes, it seems extremely important to investigate in more depth the mechanisms that may be involved in CM and MO. Calcitonin gene-related peptide (CGRP) undoubtedly plays an important, though not exclusive, role in the generation of migraine headaches. CGRP receptors are localized in the sites involved in migraine pathogenesis. CGRP is involved in mast cell degranulation, neurogenic inflammation, and vasodilation. It has been shown that CGRP induces InterLeukin-6 (IL-6) gene expression in macrophages by upregulation of circular RNA_007893, a modulator of MicroRNA-485-5p. MicroRNAs (miRNAs) are involved in the generation and maintenance of chronic pain and several lines of evidence suggest that specific miRNAs may play a role in migraine pain. In a previous clinical study, Andersen and colleagues found an increased expression of miR-34a-5p during migraine attacks, while miR-382-5p levels increased also in the attack-free phase. In addition, the peripheral expression of miR-34a-5p decreased in the saliva of young migraineurs patients under drug treatment, thus suggesting a possible role in the prediction of therapeutic response. At present, no reliable individual biomarker of migraine and its subtypes has been identified, though multiple molecules have been proposed and supported by promising results.

In this study, the investigators assayed the plasma levels of CGRP and the expression of miRNAs in PBMCs of patients with EM and CM-MO in order to identify individual or a panel of potential biomarkers of migraine subtypes. As secondary outcome, the investigators evaluated the changes in CGRP and miRNAs levels after detoxification in the subjects with CM-MO in order to gather more insights into the mechanisms that are involved in the improvement of migraine pattern following the withdrawal of the overused medications.

This is a cross-sectional observational controlled study with 2 groups (EM and CM-MO), integrated with a prospective open label interventional trial to assess the effect of detoxification in the CM-MO group on the biomarkers of interest. Samples were labeled with numerical codes and all biochemical determinations were performed by researchers who were blind to the diagnosis.

At baseline (Day 0), all patients underwent a visit with a neurologist of the Headache Science Centre during which clinical/demographical data were recorded and inclusion/exclusion criteria were checked. If the criteria were met, subjects underwent peripheral venipuncture for the evaluation of CGRP, miR-382-5p, and miR-34a-5p levels.

Patients with CM-MO were hospitalized for a 7-day standardized detoxification protocol, consisting in abrupt withdrawal of overused drugs associated to intravenous therapy twice daily (08:00 a.m. and 4:00 p.m.) with isotonic 0.9% Sodium Chloride (NaCl) saline 500 ml + cyanocobalamin 2500 mcg + folic acid 0.70 mg + nicotinamide 12 mg + ascorbic acid 150 mg + sodic glutathione 600 mg + delorazepam 0.5 mg. Two months after hospital discharge (Day 1), the CM-MO patients returned for a follow-up visit, during which clinical data were recorded and a second venous blood sample obtained from their ante-cubital vein.

ELIGIBILITY:
Inclusion Criteria for EM subjects:

* diagnosis of migraine without aura according to The International Classification Headache Disorders 3rd edition (ICHD-3) criteria;
* documented history of EM for at least 10 years before enrollment;
* negative life-time history of CM.

Exclusion Criteria:

* headache or headache with migraine features and mild intensity (less than 4 on 0 to 10 visual analogue scale) in the 24 hours before blood sampling;
* intake of acute anti-migraine medications in the 24 hours before blood sampling.

Inclusion criteria for CM-MO patients:

* diagnosis of CM and MO according to ICHD-3 criteria;
* documented pattern of stable CM in the 5 years prior to enrollment, without any remission period. This latter point was verified with a high degree of confidence combining the information obtained from the patients' history with their medical records, including their headache diaries.

Exclusion Criteria:

* headache or headache with migraine features and mild intensity (less than 4 on 0 to 10 visual analogue scale) in the 24 hours before blood sampling;
* intake of acute anti-migraine medications in the 24 hours before blood sampling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty-seven subjects with EM and 28 subjects with CM-MO were consecutively enrolled among patients attending the outpatient clinics of the Headache Science Centre of the IRCCS Mondino Foundation of Pavia (Italy).
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Plasma levels of CGRP | Day 0 at the enrolment
  In order to identify individual or a panel of potential biomarkers of migraine subtypes
Expression of miRNAs in PBMCs | Day 0 at the enrolment
  In order to identify individual or a panel of potential biomarkers of migraine subtypes

SECONDARY OUTCOMES:
Changes in CGRP levels | Day1 - Two months after Day 0
  In the subjects with CM-MO after detoxification in order to gather more insights into the mechanisms that are involved in the improvement of migraine pattern following the withdrawal of the overused medications.
Changes in miRNAs levels | Day 1 - Two months after Day 0
  In the subjects with CM-MO after detoxification in order to gather more insights into the mechanisms that are involved in the improvement of migraine pattern following the withdrawal of the overused medications.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, Prof, Principal Investigator — IRCCS Mondino Foundation, Pavia
Locations (1):
- Headache Science Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diener HC, Tassorelli C, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ, Mandrekar J; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of acute treatment of migraine attacks in adults: Fourth edition. Cephalalgia. 2019 May;39(6):687-710. doi: 10.1177/0333102419828967. Epub 2019 Feb 26. PMID 30806518
- [Background] Xu J, Kong F, Buse DC. Predictors of episodic migraine transformation to chronic migraine: A systematic review and meta-analysis of observational cohort studies. Cephalalgia. 2020 Apr;40(5):503-516. doi: 10.1177/0333102419883355. Epub 2019 Oct 21. PMID 31635478
- [Background] Serrano D, Lipton RB, Scher AI, Reed ML, Stewart WBF, Adams AM, Buse DC. Fluctuations in episodic and chronic migraine status over the course of 1 year: implications for diagnosis, treatment and clinical trial design. J Headache Pain. 2017 Oct 4;18(1):101. doi: 10.1186/s10194-017-0787-1. PMID 28980171
- [Background] Tassorelli C, Jensen R, Allena M, De Icco R, Sances G, Katsarava Z, Lainez M, Leston J, Fadic R, Spadafora S, Pagani M, Nappi G; the COMOESTAS Consortium. A consensus protocol for the management of medication-overuse headache: Evaluation in a multicentric, multinational study. Cephalalgia. 2014 Aug;34(9):645-655. doi: 10.1177/0333102414521508. Epub 2014 Feb 20. PMID 24558185
- [Background] Rossi P, Faroni JV, Tassorelli C, Nappi G. Advice alone versus structured detoxification programmes for complicated medication overuse headache (MOH): a prospective, randomized, open-label trial. J Headache Pain. 2013 Feb 8;14(1):10. doi: 10.1186/1129-2377-14-10. PMID 23565591
- [Background] Meng ID, Dodick D, Ossipov MH, Porreca F. Pathophysiology of medication overuse headache: insights and hypotheses from preclinical studies. Cephalalgia. 2011 May;31(7):851-60. doi: 10.1177/0333102411402367. Epub 2011 Mar 28. PMID 21444643
- [Background] Diener HC, Dodick D, Evers S, Holle D, Jensen RH, Lipton RB, Porreca F, Silberstein S, Schwedt T. Pathophysiology, prevention, and treatment of medication overuse headache. Lancet Neurol. 2019 Sep;18(9):891-902. doi: 10.1016/S1474-4422(19)30146-2. Epub 2019 Jun 4. PMID 31174999
- [Background] De Felice M, Ossipov MH, Porreca F. Persistent medication-induced neural adaptations, descending facilitation, and medication overuse headache. Curr Opin Neurol. 2011 Jun;24(3):193-6. doi: 10.1097/WCO.0b013e328346af25. PMID 21467931
- [Background] Munksgaard SB, Bendtsen L, Jensen RH. Modulation of central sensitisation by detoxification in MOH: results of a 12-month detoxification study. Cephalalgia. 2013 May;33(7):444-53. doi: 10.1177/0333102412475235. Epub 2013 Feb 21. PMID 23431023
- [Background] De Felice M, Ossipov MH, Wang R, Lai J, Chichorro J, Meng I, Dodick DW, Vanderah TW, Dussor G, Porreca F. Triptan-induced latent sensitization: a possible basis for medication overuse headache. Ann Neurol. 2010 Mar;67(3):325-37. doi: 10.1002/ana.21897. PMID 20373344
- [Background] Lambru G, Andreou AP, Guglielmetti M, Martelletti P. Emerging drugs for migraine treatment: an update. Expert Opin Emerg Drugs. 2018 Dec;23(4):301-318. doi: 10.1080/14728214.2018.1552939. Epub 2018 Nov 30. PMID 30484333
- [Background] Deng T, Yang L, Zheng Z, Li Y, Ren W, Wu C, Guo L. Calcitonin gene-related peptide induces IL-6 expression in RAW264.7 macrophages mediated by mmu_circRNA_007893. Mol Med Rep. 2017 Dec;16(6):9367-9374. doi: 10.3892/mmr.2017.7779. Epub 2017 Oct 12. PMID 29039515
- [Background] Gallelli L, Siniscalchi A, Carotenuto M, Caroleo MC, Cione E, Guidetti V. microRNAs-based Predictor Factor in Patients with Migraine-ischemic Stroke. Microrna. 2017;6(1):17-21. doi: 10.2174/2211536606666170104130101. PMID 28056747
- [Background] Ferroni P, Barbanti P, Spila A, Fratangeli F, Aurilia C, Fofi L, Egeo G, Guadagni F. Circulating Biomarkers in Migraine: New Opportunities for Precision Medicine. Curr Med Chem. 2019;26(34):6191-6206. doi: 10.2174/0929867325666180622122938. PMID 29932027
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Cernuda-Morollon E, Larrosa D, Ramon C, Vega J, Martinez-Camblor P, Pascual J. Interictal increase of CGRP levels in peripheral blood as a biomarker for chronic migraine. Neurology. 2013 Oct 1;81(14):1191-6. doi: 10.1212/WNL.0b013e3182a6cb72. Epub 2013 Aug 23. PMID 23975872
- [Background] Andersen HH, Duroux M, Gazerani P. Serum MicroRNA Signatures in Migraineurs During Attacks and in Pain-Free Periods. Mol Neurobiol. 2016 Apr;53(3):1494-1500. doi: 10.1007/s12035-015-9106-5. Epub 2015 Feb 1. PMID 25636687
- [Background] Tassorelli C, Diener HC, Dodick DW, Silberstein SD, Lipton RB, Ashina M, Becker WJ, Ferrari MD, Goadsby PJ, Pozo-Rosich P, Wang SJ; International Headache Society Clinical Trials Standing Committee. Guidelines of the International Headache Society for controlled trials of preventive treatment of chronic migraine in adults. Cephalalgia. 2018 Apr;38(5):815-832. doi: 10.1177/0333102418758283. Epub 2018 Mar 4. PMID 29504482
- [Background] Russo AF. Calcitonin gene-related peptide (CGRP): a new target for migraine. Annu Rev Pharmacol Toxicol. 2015;55:533-52. doi: 10.1146/annurev-pharmtox-010814-124701. Epub 2014 Oct 8. PMID 25340934
- [Background] Andersen HH, Duroux M, Gazerani P. MicroRNAs as modulators and biomarkers of inflammatory and neuropathic pain conditions. Neurobiol Dis. 2014 Nov;71:159-68. doi: 10.1016/j.nbd.2014.08.003. Epub 2014 Aug 10. PMID 25119878
- [Background] Li MD, van der Vaart AD. MicroRNAs in addiction: adaptation's middlemen? Mol Psychiatry. 2011 Dec;16(12):1159-68. doi: 10.1038/mp.2011.58. Epub 2011 May 24. PMID 21606928
- [Background] Lee MJ, Lee SY, Cho S, Kang ES, Chung CS. Feasibility of serum CGRP measurement as a biomarker of chronic migraine: a critical reappraisal. J Headache Pain. 2018 Jul 13;19(1):53. doi: 10.1186/s10194-018-0883-x. PMID 30006780
- [Background] Munksgaard SB, Ertsey C, Frandsen E, Bendtsen L, Tekes K, Jensen RH. Circulating nociceptin and CGRP in medication-overuse headache. Acta Neurol Scand. 2019 Mar;139(3):269-275. doi: 10.1111/ane.13053. Epub 2018 Dec 11. PMID 30457160
- [Background] Fan PC, Kuo PH, Lee MT, Chang SH, Chiou LC. Plasma Calcitonin Gene-Related Peptide: A Potential Biomarker for Diagnosis and Therapeutic Responses in Pediatric Migraine. Front Neurol. 2019 Jan 24;10:10. doi: 10.3389/fneur.2019.00010. eCollection 2019. PMID 30733702
- [Background] Frederiksen SD, Bekker-Nielsen Dunbar M, Snoer AH, Deen M, Edvinsson L. Serotonin and Neuropeptides in Blood From Episodic and Chronic Migraine and Cluster Headache Patients in Case-Control and Case-Crossover Settings: A Systematic Review and Meta-Analysis. Headache. 2020 Jun;60(6):1132-1164. doi: 10.1111/head.13802. Epub 2020 Apr 15. PMID 32293721
- [Derived] Greco R, De Icco R, Demartini C, Zanaboni AM, Tumelero E, Sances G, Allena M, Tassorelli C. Plasma levels of CGRP and expression of specific microRNAs in blood cells of episodic and chronic migraine subjects: towards the identification of a panel of peripheral biomarkers of migraine? J Headache Pain. 2020 Oct 16;21(1):122. doi: 10.1186/s10194-020-01189-0. PMID 33066724